CLINICAL TRIAL: NCT05322005
Title: A Non-randomized Multicentre Study for the Evaluation of the Clinical Performance and Safety of the Augmentation-to-surgery and Conservative Treatments for the Degenerative Meniscopathy, With Injection of Polynucleotide Gel
Brief Title: Study of Clinical Performance and Safety of Treatments in Degenerative Meniscopathy With Injection of Polynucleotides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mastelli S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDM22M
Record Dates: First submitted 2022-03-11; First posted 2022-04-11 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Meniscus Tear; Meniscus Lesion

STUDY DESIGN:
Intervention Model Description: Treatment A (augmentation-to-surgery): subjects surgically treated with partial meniscectomy combined with an intraarticular and intra-meniscal injection of polynucleotide gel.
  Treatment B (conservative): subjects treated with three injections session of polynucleotide gel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: augmentation to surgery (Experimental): Patients will be surgically treated with partial meniscectomy combined with an intraarticular and intra-meniscal injection of polynucleotide gel, during an arthroscopic procedure. After 6 weeks the patients attend a second injection session, during an ambulatorial visit. At 8 weeks from the surgery the patients attend the third ambulatorial injection session
  Interventions: Procedure: partial meniscectomy; Device: Condrotide® (polynucleotides gel: class III medical device)
- Arm B: conservative treatment (Experimental): The patients are going to receive three injections session (polynucleotide gel) performed with a time interval of 2 weeks.
  Interventions: Device: Condrotide® (polynucleotides gel: class III medical device)

INTERVENTIONS:
Procedure: partial meniscectomy — Arthroscopic procedure
  Arms: Arm A: augmentation to surgery
Device: Condrotide® (polynucleotides gel: class III medical device) — Condrotide® Polynucleotide gel is a joint lubricating and viscosizing agent, given by intraarticular and intra-meniscal injection

SUMMARY:
This is a non-randomized multicentre study for the evaluation of the clinical performance and safaty of the augmentation-to-surgery and conservative treatments for the degenerative meniscopathies, with injection of polynucleotide gel.

DETAILED DESCRIPTION:
Meniscal tear plays a significant role among the multitude of ethiologies of knee pain. In the setting of chronic meniscus degeneration, healing potential remains low due to a vascular penetration of less than one-third of the adult meniscus. Currently, both conservative and surgical modalities can be utilized in the treatment of the painful degenerative menisci, and no gold standard treatment has been identified. Polynucleotide gel Condrotide® is a polynucleotide solution, used in case of degenerative painful join pathologies, favouring the physiological mechanism of joint repair because of the capacity to normalize the viscosity of synovial fluid and supposed to improve the joint trophism. The present study aims at evaluating the capacity of the polynucleotide gel injection to stimulate healing and slow down progression of meniscal degeneration, through augmentation-to-surgery and conservative treatments for the degenerative meniscopathies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with age between 18 and 65 years
2. Presence of symptomatic degenerative meniscus tear
3. Presence of one of the following unilateral symptoms: pain, catching, or locking of the knee
4. Non responsive to physical therapy for at least 3-4 weeks
5. Be in neutral alignment +/- 5 degrees of the mechanical axis
6. Subject must be physically and mentally willing and able to comply with the study follow-up schedule
7. Subject must sign Ethic committe approved informed consent
8. Subject is willing and able to comply with all study procedures, including visits and diagnostic procedures

Exclusion Criteria:

1. Radiographic osteoarthritis of the knee in any compartment greater than Kellgren-Lawrence (KL) grade 3.
2. Presence of bone marrow edema (BME) at the index knee.
3. Presence of knee instability.
4. Have a varus or valgus knee deformity > 5 degrees.
5. Have meniscal roots tears.
6. Have discoid meniscus.
7. Have patella instability or non-anatomically positioned patella.
8. Have a knee flexion contracture > 10 degrees.
9. Be unable to flex the knee to 90 degrees.
10. Have a leg length discrepancy causing a noticeable limp.
11. Have an active infection or tumor.
12. Have any type of knee joint inflammatory disease including Sjogren's syndrome.
13. Have neuropathic knee osteoarthropathy, also known as Charcot joint.
14. Any disorder or impairment that would interfere with evaluation of outcomes measures, such as neurological, degenerative muscular, psychiatric or cognitive conditions.
15. Participation to another clinical trial or clinical investigation in the previous 3 months.
16. BMI > 35.
17. Prior knee arthroscopy within 6 months of study enrolment.
18. Unable to have an MRI scan.
19. Known allergy, sensitivity or intolerance to any of the components of the investigational device or to products originating from fish.
20. Positive history of human immunodeficiency virus antibodies, hepatitis B surface antigen or hepatitis C virus antibodies.
21. Autoimmune diseases, rheumatoid disease eg. Lupus erythematosus.
22. The subject is currently being treated with radiation and or chemotherapy.
23. Previous or ongoing alcohol abuse or dependence, use of illicit drugs within 1 year prior to enrolment.
24. Patients who are pregnant or planning to become pregnant during the planned period of participation in the study or who are breastfeeding. Women of child-bearing age must consent to use and actually make use of a highly effective contraceptive method, considered acceptable by the investigator, for the whole study duration.
25. Does not agree to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
Overall Knee Injury Osteoarthritis Outcome Score (KOOS) will be measured | 24 months (end of follow up)
  The change of overall KOOS score will be evaluated from baseline (V1) to 6 (V6), 12 (V7), and 24 (V8) months after treatment completion.
  An improvement of 10 points in the score will be considered success.
  The KOOS score assesses; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.

SECONDARY OUTCOMES:
The change of the radiological assessment of the cartilage by a 5-points Likert scale | 24 months
  Likert scale scoring: 0=worsened; 1= not worsened or improved; 2= slightly improved; 3= improved; 4= very much improved). The articular cartilage and meniscal appearance change will be evaluated from baseline (V1) to 6 (V6), 12 (V7), 24 (V8) months after treatment completion (T0).
The change of the International Knee Documentation Committee (IKDC Questionnaire) | 24 months
  Is a knee-specific patient-reported outcome measure. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
The change of the Tegner activity score from baseline (V1) to 3 (V5), 6 (V6), 12 (V7), 24 (V8) months after treatment completion (T0). | 24 months
  The Tegner activity scale is a one-item score evaluating work and sports activities on a scale of 0 to 10. Zero represents disability.
AE and device deficiencies Reporting | 24 months
  Will be evaluated:
  * number and typology of device- or procedure-related serious adverse events (SAEs)
  * the number and typology of all other adverse events (AEs) or SAEs;
  * the number and typology of device deficiencies (DD)

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, Prof., Principal Investigator — Plastic surgery IRCCS Humanitas; Peter Verdonk, Prof., Principal Investigator — Monica Ziekenhuizen Antwerpen en Deurne
Locations (2):
- Peter Verdonk, Deurne, Belgium
- Elizaveta Kon, Milan, Milan, Italy